CLINICAL TRIAL: NCT03788018
Title: Effect of Intravenous Lidocaine Combined With Dexmedetomidine on Postoperative Nausea and Vomiting After Laparoscopic Hysterectomy
Brief Title: Effect of Lidocaine Plus Dexmedetomidine Infusion on PONV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Siqi (Other)
Responsible Party: Sponsor-Investigator, Xu Siqi, Department of Anesthesiology, Anqing Municipal Hospital
Organization: Anqing Municipal Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AnqingMH
Record Dates: First submitted 2018-12-20; First posted 2018-12-27 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Lidocaine; Dexmedetomidine; Nausea and Vomiting, Postoperative
Keywords: Lidocaine; Dexmedetomidine; Postoperative nausea and vomiting; laparoscopic hysterectomy
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Effect of IV lidocaine and dexmedetomidine on PONV (Experimental)
  Interventions: Drug: lidocaine and dexmedetomidine IV; Drug: saline IV
- Effect of IV saline on PONV (Experimental)
  Interventions: Drug: lidocaine and dexmedetomidine IV; Drug: saline IV

INTERVENTIONS:
Drug: lidocaine and dexmedetomidine IV — Patients received IV bolus infusion of lidocaine (2%) 1.5 mg/kg and dexmedetomidine 0.5 µg/kg diluted with normal saline to 20 ml in the LD group respectively, over 10 minutes before induction of anesthesia, followed by a continuous IV infusion at rate of lidocaine 1.5 mg/kg and dexmedetomidine 0.4 µg/kg made up to 20 mL every hour until 30 min before the end of operation, respectively.
Drug: saline IV — Patients received 20 ml normal saline and 20 ml normal saline in the CON group respectively, over 10 minutes before induction of anesthesia, followed by a continuous IV infusion 20 ml normal saline and 20 ml normal saline every hour until 30 min before the end of surgery

SUMMARY:
BACKGROUND: Few researches have manifested that intravenous (IV) lidocaine or dexmedetomidine decreased the incidence of postoperative nausea and vomiting (PONV). The investigators investigated whether IV lidocaine plus dexmedetomidine infusion could better reduce the incidence of PONV after laparoscopic hysterectomy.

METHODS: One hundred and twenty women with elective laparoscopic hysterectomy were randomly divided into two groups: patients in the lidocaine combined with dexmedetomidine group (LD group, n=60) received lidocaine (1.5 mg/kg loading, 1.5 mg/kg/h infusion) and dexmedetomidine (0.5 μg/kg loading, 0.4 μg/kg/h infusion) respectively. Patients in the control group (CON group, n=60) received the equal volume of saline. Primary outcome was the incidence of the first 48 h nausea, vomiting and PONV after surgery. The secondary outcomes included perioperative propofol and remifentanil consumption, postoperative fentanyl requirement, Ramsay sedation score, and bradycardia during post-anaesthesia care unit (PACU) stay.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical statusⅠand Ⅱ
* Aged 40-55 years
* Scheduled for elective laparoscopic hysterectomy

Exclusion Criteria:

* History of allergy to local anesthetics
* Severe respiratory disease
* Renal or hepatic insufficiency
* History of preoperative opioids medication and psychiatric
* preoperative bradycardia
* preoperative atrioventricular block
* Subjects who experienced severe hypotension (mean arterial pressure [MAP] <60 mmHg) or bradycardia (heart rate [HR] <40 bpm), urticaria, or arrhythmia during lidocaine and dexmedetomidine infusion period

Ages: 40 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-11-15 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
postoperative nausea | 0-2 hours after surgery
  Our primary outcome was the incidence of nausea during the 0-2 hours after surgery
postoperative nausea | 2-24 hours after surgery
  Our primary outcome was the incidence of nausea during the 2-24 hours after surgery
postoperative nausea | 24-48 hours after surgery
  Our primary outcome was the incidence of nausea during the 24-48 hours after surgery
postoperative vomiting | 0-2 hours after surgery
  Our primary outcome was the incidence of vomiting during the 0-2 hours after surgery
postoperative vomiting | 2-24 hours after surgery
  Our primary outcome was the incidence of vomiting during the 2-24 hours after surgery
postoperative vomiting | 24-48 hours after surgery
  Our primary outcome was the incidence of vomiting during the 24-48 hours after surgery
postoperative nausea and vomiting (PONV) | 0-2 hours after surgery
  Our primary outcome was the incidence of PONV during the 0-2 hours after surgery
postoperative nausea and vomiting (PONV) | 2-24 hours after surgery
  Our primary outcome was the incidence of PONV during the 2-24 hours after surgery
postoperative nausea and vomiting (PONV) | 24-48 hours after surgery
  Our primary outcome was the incidence of PONV during the 24-48 hours after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anqing Hospital Anesthesiology, Anqing, Anhui, China

IPD SHARING:
Plan to Share IPD: No